CLINICAL TRIAL: NCT04309695
Title: The Zenflow Spring System Safety and Performance Study (ZEST CAN)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zenflow, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0111
Record Dates: First submitted 2020-03-04; First posted 2020-03-16 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2020-08

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Receives intervention with the Zenflow Spring System.
  Interventions: Device: Zenflow Spring System

INTERVENTIONS:
Device: Zenflow Spring System — The Zenflow Spring is a nitinol urethral implant for the treatment of Lower Urinary Tract Symptoms (LUTS) that arise due to bladder outlet obstruction (BOO), secondary to the presence of Benign Prostatic Hypertrophy (BPH). The device is intended to be a permanent implant however it may be removed if necessary.

SUMMARY:
The objectives of the trial are to demonstrate the safety and performance of the Zenflow Spring System in relieving the symptoms of obstructive Benign Prostatic Hyperplasia (BPH).

DETAILED DESCRIPTION:
The purpose of the Zenflow Study (ZEST CAN) is to evaluate the safety, performance and effectiveness of the Zenflow Spring System for the treatment of Lower Urinary Tract Symptoms (LUTS) that arise due to bladder outlet obstruction (BOO), secondary to the presence of Benign Prostatic Hyperplasia (BPH). It is intended that the features of the Zenflow Spring will provide an effective office-based treatment and management therapy for BPH with little or no side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able and willing to comply with all the assessments of the study
2. Patient or patient's legal representative has been informed of the nature of the study, agrees to participate and has signed the informed consent form
3. ≥ 45 years of age
4. Baseline IPSS score > 13
5. Prostate volume 25 - 80 cc and prostatic urethral length between 2.5-4.5 cm measured within the past 90 days
6. Failed, intolerant, or patient choice to not take a medication regimen for the treatment of LUTS

Exclusion Criteria:

1. Obstructive intravesical median prostatic lobe which in the opinion of the operator would not benefit from treatment
2. Urethral stricture, meatal stenosis, or bladder neck obstruction - either current, or recurrent requiring 2 or more dilations as reported in the patient's history
3. Requiring self-catheterization to void.
4. Baseline PSA > 10 ng/mL or confirmed or suspected prostate cancer
5. Any of the following, taken from a single uroflowmetry reading:

   1. Post-void residual volume (PVR) > 250 ml
   2. Peak urinary flow rate of > 15 ml/second
   3. < 125 ml urinary volume voided at baseline (pre-bladder urinary volume of ≥150 ml required)
6. Other condition or disease that might cause urinary retention
7. History of other diseases causing voiding dysfunction
8. Concomitant Urinary Tract Infection (UTI) (subject can be enrolled following successful treatment of UTI and a clean urine test), or subjects who have a history of recurrent or chronic UTIs (defined as 2 or more UTIs in the past 12 months)
9. Concomitant bladder stones
10. Previous pelvic irradiation or radical pelvic surgery
11. Previous prostate surgery, stent implantations, laser prostatectomy, hyperthermia or another invasive treatment to the prostate
12. Chronic prostatitis, or recurring prostatitis within the past 12 months
13. Known allergy to nickel
14. Life expectancy less than 24 months
15. Use of concomitant medications (e.g., anticholinergics, antispasmodics or tricyclic antidepressants) affecting bladder function
16. Inability to stop taking anticoagulants and/or antiplatelets for at least 3 days prior to the procedure or coumadin for at least 5 days prior to the procedure (low dose aspirin therapy not prohibited).
17. Taking 5-alpha-reductase inhibitors within 3 months of pre-treatment (baseline) evaluation
18. Taking one of the following within 2 weeks of pre-treatment (baseline) evaluation:

    1. alpha-blockers,
    2. imipramine,
    3. anticholinergics, or
    4. cholinergic medication gonadotropin releasing hormonal analogs
19. Taking androgens, unless evidence of eugonadal state for at least 6 months.
20. Taking one of the following within 24 hours of pre-treatment (baseline) evaluation:

    1. phenylephrine, or
    2. pseudoephedrine
21. Future fertility concerns
22. Any concurrent medical condition or illness that might prevent study completion or would confound study results

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Successful placement of the Zenflow Spring Implant | Day of discharge up to 7 days following device placement
  Number of successful deployments and procedural successes for the Zenflow System to implant the Spring device in the OR, or in an out-patient clinical setting as compared to total treatment attempts.
Effectiveness of the Spring Implant in reducing symptoms of Benign Prostatic Hyperplasia (BPH) using the International Prostate Symptom Score | 3 month
  At 3 months, achieve at least 30% mean improvement in International Prostate Symptom Score (IPSS) compared to baseline. The patient is asked to respond to 7 questions related to his urinary health using a rating scale of 0 to 5 where zero is excellent and 5 is the worst possible. The responses to the 7 questions are tallied for a total IPSS score.
Need for urinary catheterization | 7 days after the procedure
  Achieve < 12% rate of extended post-operative urinary catheterization, defined as an occurrence of a subject requiring catheterization within the first 3 days as part of a postoperative management for inability to void, for greater than 7 days.
Incidence of procedure or device related serious adverse events | 30 days after the procedure
  Achieve < 12% rate of device or procedure related SAEs through discharge and 30 days follow up.

SECONDARY OUTCOMES:
Assessment of Sexual Health Assessment: Change in sexual health measured by change in the Sexual Health Inventory for Men (SHIM) questionnaire score | Baseline, 3, 6, 12, 24, 36, 48, & 60 months
  The patient selects the most appropriate response to 5 questions about his sexual health. Each response has an assigned value between 1 and 5. The numeric values are tallied for a total score.
Assessment of Pain, evaluated using a Visual Analog Score (VAS) of 1 to 10 | Baseline, interoperative (if conscious sedation used), immediately post-treatment, 2 weeks, 1 and 3 months
  Patient describes pain on a Visual Analog Scale (VAS). The scale is a line labeled 1 at the far left indicating minimal pain and 10 on the right, which is maximum pain.
Assessment of Adverse Events | Up to 5 years
  Rate of adverse events related to the procedure or device.
Assessment of Clavien-Dindo events | Up to 5 years
  Proportion of subjects with procedure or device related adverse events classified as Clavien-Dindo Grade 3 or higher or any event resulting in persistent disability evidenced through 3 months post treatment.
Assessment of PSA | Up to 5 years
  Change in PSA from baseline through 12, 24, 36, 48, & 60 months post treatment.
Effectiveness of the Spring Implant in reducing symptoms of Benign Prostatic Hyperplasia (BPH) | Baseline, 2 weeks, 1, 6, 12, 24, 36, 48, & 60 months
  The patient is asked to respond to 7 questions related to his urinary health using a rating scale of 0 to 5 where zero is excellent and 5 is the worst possible. The responses to the 7 questions are tallied for a total score
Effectiveness of the Spring Implant in reducing symptoms of Benign Prostatic Hyperplasia (BPH) | Baseline, 2 weeks, 1, 3, 6, 12, 24, 36, 48, & 60 months
  Improvement in flow of urine as measured by uroflowmetry machine.
Effectiveness of the Spring Implant in reducing symptoms of Benign Prostatic Hyperplasia (BPH) | Up to 5 years
  Incidence of increase in dosage or initiation of new medication to treat symptoms of BPH.
Effectiveness of the Spring Implant in reducing symptoms of Benign Prostatic Hyperplasia (BPH) | 24 to 60 months
  Incidence of repeat treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Toronto Western Hospital, Toronto, Ontario
  - Groupe Sante Brunswick, Pointe-Claire, Quebec

IPD SHARING:
Plan to Share IPD: No